CLINICAL TRIAL: NCT01279681
Title: Randomized Phase III Trial of mFOLFOX7 or XELOX Plus Bevacizumab Versus 5-Fluorouracil/Leucovorin or Capecitabine Plus Bevacizumab as First-line Treatment in Elderly Patients With Metastatic Colorectal Cancer
Brief Title: Combination Chemotherapy Plus Bevacizumab With or Without Oxaliplatin in Treating Older Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N0949; NCCTG-N0949; CDR0000692257 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-02622 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-11

CONDITIONS: Cognitive/Functional Effects; Colorectal Cancer; Neurotoxicity
Keywords: neurotoxicity; cognitive/functional effects; stage IVA colon cancer; stage IVA rectal cancer; stage IVB colon cancer; stage IVB rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neurotoxicity Syndromes; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Capecitabine; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A [fluoropyrimidine + bevacizumab (BEV)] (Active Comparator): Patients receive either 5FU/LV or Capecitabine, plus BEV. 5FU/LV + BEV is comprised of 5FU IV over 46-48 hours, LV calcium IV over 2 hours, and BEV IV over 10-90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. Capecitabine + BEV is comprised of capecitabine PO BID on days 1-14 and BEV IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: capecitabine; Drug: fluorouracil; Drug: leucovorin calcium
- Arm B [fluoropyrimidine/oxaliplatin (OXAL) + BEV] (Experimental): Patients receive either mFOLFOX7 plus BEV, or Capecitabine + OXAL (XELOX) plus BEV. mFOLFOX7 + BEV is comprised of OXAL IV over 2 hours, LV calcium IV over 2 hours, and 5FU IV over 46-48 hours on day 1. Patients also receive BEV IV over 10-90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. XELOX + BEV is comprised of OXAL IV over 2 hours on day 1 and capecitabine PO BID on days 1-14. Patients also receive BEV IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: capecitabine; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin

INTERVENTIONS:
Biological: bevacizumab — Given IV
Drug: capecitabine — Given PO
Drug: fluorouracil — Given IV
Drug: leucovorin calcium — Given IV
Drug: oxaliplatin — Given IV
  Arms: Arm B [fluoropyrimidine/oxaliplatin (OXAL) + BEV]

SUMMARY:
This randomized phase III trial studies how well combination chemotherapy plus bevacizumab with or without oxaliplatin works in treating older patients with colorectal cancer that has spread to other places in the body. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Monoclonal antibodies, such as bevacizumab, may block tumor growth in different ways by targeting certain cells. Bevacizumab may also stop the growth of cancer by blocking blood flow to the tumor. It is not yet known whether combination chemotherapy plus bevacizumab is more effective with or without oxaliplatin in treating colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the progression-free survival (PFS) of elderly patients with metastatic colorectal carcinoma who are randomized to receive fluoropyrimidine (fluorouracil)-based therapy plus bevacizumab, with or without oxaliplatin.

SECONDARY OBJECTIVES:

I. In a prospectively planned pooled analysis with a similar trial to be conducted by the Japanese Clinical Oncology Group (JCOG), evaluate and compare the overall survival (OS) of elderly patients with metastatic colorectal carcinoma who are randomized to receive fluoropyrimidine-based therapy plus bevacizumab, with or without oxaliplatin.

II. To assess and compare response rates and adverse events of elderly patients with metastatic colorectal carcinoma randomized to receive fluoropyrimidine-based therapy plus bevacizumab, with or without oxaliplatin.

OUTLINE: Patients are randomized to 1 of 2 treatment arms and assigned to treatment groups based on physician decision for fluoropyrimidine.

ARM A: Patients receive either 5FU/LV or Capecitabine, plus BEV. 5FU/LV + BEV is comprised of 5FU IV over 46-48 hours, LV calcium IV over 2 hours, and BEV IV over 10-90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. Capecitabine + BEV is comprised of capecitabine PO BID on days 1-14 and BEV IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive either mFOLFOX7 plus BEV, or Capecitabine + OXAL (XELOX) plus BEV. mFOLFOX7 + BEV is comprised of OXAL IV over 2 hours, LV calcium IV over 2 hours, and 5FU IV over 46-48 hours on day 1. Patients also receive BEV IV over 10-90 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. XELOX + BEV is comprised of OXAL IV over 2 hours on day 1 and capecitabine PO BID on days 1-14. Patients also receive BEV IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria

* Patients must have metastatic colorectal cancer that has been histologically or cytologically confirmed; Note: histologic confirmation can be obtained from the primary tumor with appropriate imaging studies confirming metastatic spread
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Peripheral platelet count (PLT) >= 100,000/mm^3
* Hemoglobin (HgB) > 9.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate transaminase (AST) =< 2.5 x ULN (=< 5 x ULN for patients with liver involvement)
* Alkaline phosphatase =< 3 x ULN (=< 5 x ULN for patients with liver involvement)
* Creatinine =< 1.5 x ULN
* International normalized ratio (INR) < 1.5 x ULN unless patients are receiving anti-coagulation therapy; patients receiving prophylactic anti-coagulation therapy with an agent such as warfarin or heparin are allowed to participate if INR =< 3.0
* Urine protein creatinine (UPC) ratio < 1 or urine dipstick < 2+

  * NOTE: Urine protein must be screened by urine analysis for urine protein creatinine (UPC) ratio or by dip stick; for UPC ratio >= 1.0 or urine dipstick >= 2+, 24-hour urine protein must be obtained and the level should be < 1000 mg
* Life expectancy >= 3 months
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide informed written consent
* Willing to provide mandatory blood samples for correlative research purposes

Exclusion Criteria

* Men of child bearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of the safety and adverse events of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticoid steroids) including patients known to be human immunodeficiency virus (HIV) positive with cluster of differentiation (CD)4 < 100 cells/uL
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 3 years prior to randomization; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history of prior malignancy, patients must not be receiving other specific treatment (other than hormonal therapy) for this prior cancer
* Prior chemotherapy, radiation therapy, immunotherapy, or biological therapy for recurrent or metastatic colorectal cancer

  * NOTE: prior chemotherapy or radiotherapy is permitted if they had been administered as adjuvant or neoadjuvant therapy and a complete surgical resection of the original colorectal cancer had been achieved
* Progressive disease =< 12 months of completing oxaliplatin-containing adjuvant therapy
* Prior radiation to > 30% of the bone marrow at any time
* Calculated creatinine clearance < 60 mL/minute

  * NOTE: If calculated creatinine clearance does not meet eligibility requirement, a 24-hour urine can be collected for a creatinine clearance, and the patient can been rolled if measured creatinine clearance >= 60 mL/minute
* Known central nervous system or brain metastasis that are either symptomatic or untreated; Note: if a patient has a resection of the metastasis and is no longer symptomatic, the patient is eligible for the study; Note: patients with neurological symptoms must undergo a computed tomography (CT) scan/magnetic resonance imaging (MRI) of the brain to exclude brain metastasis
* New York Heart Association (NYHA) classification III or IV congestive heart failure
* Inadequately controlled hypertension (systolic blood pressure of > 150 mm Hg or diastolic blood pressure > 100 mm Hg on anti-hypertensive medications)
* Major surgical procedures, open biopsy or significant traumatic injury =< 28 days prior to randomization or anticipation of need for elective or planned major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedures =< 7 days prior to randomization

  * NOTE: Placement of a vascular access device is allowed
* Active or recent hemoptysis (>= ½ teaspoon of bright red blood per episode) =< 30 days prior to randomization
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess =< 6 months prior to randomization
* Serious non-healing wound, active ulcer, or untreated bone fracture

  * NOTE: patients with fractures secondary to metastatic disease are eligible after appropriate radiotherapy
* History of hypertensive crisis or hypertensive encephalopathy
* Patient has experienced any arterial thromboembolic events including, but not limited to myocardial infarction, stroke, transient ischemic attack (TIA), cerebrovascular accident, unstable angina =< 6 months prior to randomization or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection) or recent peripheral arterial thrombosis =< 6 months prior to randomization
* Evidence or history of bleeding diathesis (greater than normal risk of bleeding) or coagulopathy (in the absence of therapeutic anticoagulation) any hemorrhage/bleeding event > grade 3 =< 4 weeks prior to randomization; patients with full-dose anticoagulants are eligible provided the patient has been on a stable dose, at least 2 weeks, of low molecular weight heparin or warfarin and has an INR range 2-3; aspirin doses > 325 mg daily are not allowed
* Known hypersensitivity to any of the components of 5-fluorouracil/leucovorin, capecitabine, oxaliplatin, or bevacizumab
* Clinically significant peripheral neuropathy at the time of randomization (defined in the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v]4.0 as >= grade 2 neurosensory or neuromotor toxicity)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Axel Grothey, MD, Study Chair — Mayo Clinic

REFERENCES:
- [Derived] McCleary NJ, Hubbard J, Mahoney MR, Meyerhardt JA, Sargent D, Venook A, Grothey A. Challenges of conducting a prospective clinical trial for older patients: Lessons learned from NCCTG N0949 (alliance). J Geriatr Oncol. 2018 Jan;9(1):24-31. doi: 10.1016/j.jgo.2017.08.005. Epub 2017 Sep 13. PMID 28917648

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-two participants were enrolled between January 2011 and December 2012. The trial was terminated prematurely due to poor accrual and limited cooperative group resources. All follow-up was discontinued November 1, 2014.
Pre-assignment Details: Prior to randomization, physician chose fluoropyrimidine type [ie, oral Capecitabine (Xeloda) or infusional 5FU]. Patient was randomly assigned to arm A [fluoropyrimidine + bevacizumab (BEV)] or arm B [fluoropyrimidine/oxaliplatin (OXAL) + BEV] using chosen fluoropyrimidine. LV=Leucovorin, mFOLFOX7=5FU+LV+OXAL.
Period: Overall Study
Arm/Group | Arm A [Fluoropyrimidine + Bevacizumab (BEV)] | Arm B [Fluoropyrimidine/Oxaliplatin (OXAL) + BEV]
Started | 15 | 17
Completed | 0 | 0
Not Completed | 15 | 17
Not completed — Disease Progression | 9 | 6
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Adverse Event | 2 | 3
Not completed — Death | 0 | 1
Not completed — Withdrawal Prior to Beginning Treatment | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Other Reason | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A [Fluoropyrimidine + Bevacizumab (BEV)] | Arm B [Fluoropyrimidine/Oxaliplatin (OXAL) + BEV] | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Continuous [Median (Full Range); unit: years] | 75 [71 to 81] | 77 [71 to 86] | 75.5 [71 to 86]
Age, Customized [Count of Participants; unit: Participants]
  70-74 years | 7 | 7 | 14
  75-79 years | 7 | 7 | 14
  80-84 years | 1 | 2 | 3
  85+ years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 9 | 11 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13 | 17 | 30
  Black or African American | 2 | 0 | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Performance Status was defined as 0=Asymptomatic and fully active, 1=Symptomatic and fully ambulatory, 2=Symptomatic and ambulatory.
  Participants
    0-1 | 14 | 15 | 29
    2 | 1 | 2 | 3
Number of Metastatic Sites [Count of Participants; unit: Participants]
  1 | 5 | 5 | 10
  >1 | 10 | 12 | 22
Physician determined 5-FU choice prior to randomization [Count of Participants; unit: Participants]
  Infusional | 7 | 13 | 20
  Capecitabine | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Progression free survival was defined as the time (in months) from the date of randomization to the date of documented disease progression or death, whichever occurs first. Patients were followed until progression (and progression was declared) regardless of whether the patient was on the first line treatment or not. Patients who progress following a missed scan will have their date of progression back-dated to the date of missing scan. Patients without a progression who are still alive at the time of analysis will be censored at the date of last follow-up.
Time Frame: Up to 5 years
Population: One participant who refused to initiate study treatment following randomization was excluded from the analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A [Fluoropyrimidine + Bevacizumab (BEV)] | Arm B [Fluoropyrimidine/Oxaliplatin (OXAL) + BEV]
Number analyzed (Participants) | 15 | 16
months | 6.7 [5.7 to 13.4] | 6.7 [6.0 to 10.6]
Statistical Analysis 1: Comparison: Arm A [Fluoropyrimidine + Bevacizumab (BEV)] vs Arm B [Fluoropyrimidine/Oxaliplatin (OXAL) + BEV]; Test type: Superiority or Other; p = 0.93, Regression, Cox; Cox Proportional Hazard = 1.03, 95% CI 2-sided [0.49 to 2.17]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time (in months) from randomization to death.
Time Frame: Up to 5 years
Population: One participant who refused to initiate study treatment following randomization was excluded from the analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A [Fluoropyrimidine + Bevacizumab (BEV)] | Arm B [Fluoropyrimidine/Oxaliplatin (OXAL) + BEV]
Number analyzed (Participants) | 15 | 16
months | 18.8 [16.1 to 29.3] | 15.4 [9.9 to NA] — Upper limit of 95% CI is not attainable due to insufficient number of participants with events

3. Secondary Outcome: Response Rate, Defined as the Percentage of Patients in Each Arm Who Have an Objective Status of Complete Response or Partial Response, Confirmed by a Second Assessment Measured at Least 6 Weeks From the Initial Assessment
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria:
  * Complete Response (CR): disappearance of all target lesions;
  * Partial Response (PR) 30% decrease in sum of longest diameter of target lesions;
  * Progressive Disease (PD): 20% increase in sum of longest diameter of target lesions;
  * Stable Disease (SD): small changes that do not meet above criteria.
  Response rate is reported as the percentage of participants who achieved Complete Response or Partial Response.
Time Frame: Up to 5 years
Population: One participant who refused to initiate study treatment following randomization was excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A [Fluoropyrimidine + Bevacizumab (BEV)] | Arm B [Fluoropyrimidine/Oxaliplatin (OXAL) + BEV]
Number analyzed (Participants) | 15 | 16
percentage of participants | 47 [21 to 73] | 38 [15 to 65]

4. Secondary Outcome: Number of Participants With Grade 3 Adverse Events At Least Possibly Related to Treatment
Description: Adverse events were assessed using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: Up to 42 days after treatment discontinuation
Population: One participant who refused to initiate study treatment following randomization was excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A [Fluoropyrimidine + Bevacizumab (BEV)] | Arm B [Fluoropyrimidine/Oxaliplatin (OXAL) + BEV]
Number analyzed (Participants) | 15 | 16
Participants
  Palmar-plantar erythrodysesthesia | 5 | 1
  Hypertension | 2 | 4
  Thromboembolic events | 1 | 1
  Anemia | 0 | 1
  Neutropenia | 0 | 1
  Nausea | 1 | 0
  Vomiting | 0 | 1
  Mucositis | 1 | 1
  Fatigue | 2 | 1
  Peripheral sensory neuropathy | 0 | 1
  Fall | 1 | 0
  Anorexia | 2 | 0
  Hyperglycemia | 0 | 1
  Hyponatremia | 2 | 1
  Dysesthesia | 0 | 1
  Ejection fraction descreased | 0 | 1
  Chronic kidney disease | 0 | 1
  Back pain | 0 | 1

5. Other Pre Specified Outcome: Change in Geriatric/Frailty Using the North Central Cancer Treatment Group (NCCTG) Brief Frailty Inventory and the Rockwood Frailty Index Physician and Patient-reported Items
Description: The various measures of geriatric/frailty (Canadian Geriatric Society [CGSA], Rockwood, and NCCTG measures) will be compared head to head using Bland-Altman methods to assess the differences between clinician and patient reported frailty and the relative information obtained from the various assessments. This will be the first head to head comparison of its type to assess geriatric/frailty measures.
Time Frame: Baseline to 42 days after termination of study treatment
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in QOL Using the Fatigue/Uniscale Assessment, Linear Analog Self-Assessment (LASA), and the European Quality of Live Five Dimensions Questionnaire (EQ-5D)
Description: A cut-point of 5 or lower on the overall QoL question will be defined to be the primary cut-off for analysis as that has been demonstrated to represent clinically deficient QoL.
Time Frame: Baseline to up to 42 days after termination of study treatment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Proportion of Patients Reporting Satisfaction Using the Was It Worth IT (WIWI) Questionnaire
Description: WIWI will be summarized descriptively to identify the number of patients who were satisfied with each treatment and indications for improvements therein. Proportion of patients' satisfaction will be compared between treatments by a Fisher's exact test. The impact of the clinical trial on patient QOL will be summarized via means and standard deviations and compared between treatment arms via a Wilcoxon rank sum test.
Time Frame: Baseline to up to 42 days after termination of study treatment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Overall Incidence of Grade >= 3 Toxicity in Elderly Patients
Description: A logistic regression model will be used to determine the odd ratios for the occurrence of grade 3 + toxicity with a 95% confidence interval, and the overall association will be assessed by a likelihood ratio test with a two-sided alpha level of 0.05. As a secondary analysis, a multivariate logistic model will be applied including covariates for treatment arm and the stratification factors: age, PS and metastatic sites.
Time Frame: Up to 42 days after discontinuation of treatment
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Prognostic Single-nucleotide Polymorphisms (SNPs) for Grade 3+ Hypertension
Description: Logistic regression models and conditional inference trees (or more generally conditional random forests) will be used to construct multi-variable models based on the SNPs identified as interesting.
Time Frame: Up to 42 days after treatment discontinuation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Excluded one participant who refused to initiate study treatment following randomization.
Arm/Group | Arm A [Fluoropyrimidine + Bevacizumab (BEV)] | Arm B [Fluoropyrimidine/Oxaliplatin (OXAL) + BEV]
Serious Adverse Events (participants affected / at risk) | 5/15 | 3/16
Other Adverse Events (participants affected / at risk) | 15/15 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A [Fluoropyrimidine + Bevacizumab (BEV)] (N=15) | Arm B [Fluoropyrimidine/Oxaliplatin (OXAL) + BEV] (N=16)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A [Fluoropyrimidine + Bevacizumab (BEV)] (N=15) | Arm B [Fluoropyrimidine/Oxaliplatin (OXAL) + BEV] (N=16)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (6)
Abdominal pain (Gastrointestinal disorders) | 7 (13) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 11 (73) | 11 (41)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 2 (3)
Mucositis oral (Gastrointestinal disorders) | 7 (33) | 6 (14)
Nausea (Gastrointestinal disorders) | 12 (33) | 8 (31)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 7 (12) | 3 (3)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 14 (129) | 15 (106)
Fever (General disorders) | 1 (3) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 2 (4) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 2 (2)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (3)
Weight loss (Investigations) | 7 (24) | 7 (10)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 9 (44) | 8 (33)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dysesthesia (Nervous system disorders) | 3 (7) | 5 (23)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 5 (57) | 8 (32)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (77) | 9 (65)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (6) | 1 (1)
Proteinuria (Renal and urinary disorders) | 7 (22) | 4 (11)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (4)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 (24) | 1 (6)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Hypertension (Vascular disorders) | 11 (79) | 9 (48)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Thromboembolic event (Vascular disorders) | 3 (4) | 2 (2)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less